CLINICAL TRIAL: NCT01348477
Title: Comparison Between Elliptical Domed Mesh Technique and Lichtenstein Technique, to Reduce Postoperative Pain in Open Inguinal Hernia Repair
Brief Title: Comparison Between Elliptical Domed Mesh Technique and Lichtenstein Technique in Inguinal Hernia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Smolinski Kurek Rafal Ludwik, Mexican Social Security Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2010-1005-10
Record Dates: First submitted 2011-05-02; First posted 2011-05-05 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2010-09

CONDITIONS: Inguinal Hernia
Keywords: inguinal; hernia; pain; inguinodynia; mesh
MeSH Terms: conditions — Hernia, Inguinal; Hernia; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elliptical domed mesh technique (Experimental): 84 adult patients with primary uncomplicated inguinal hernia, treated with an open preperitoneal elliptical mesh technique
  Interventions: Procedure: Elliptical domed mesh technique
- Lichtenstein technique (Active Comparator): 84 adult patients with primary uncomplicated inguinal hernia treated with the Lichtenstein technique (gold standard)
  Interventions: Procedure: Elliptical domed mesh technique

INTERVENTIONS:
Procedure: Elliptical domed mesh technique — A segment of polypropylene mesh of 10 by 15cm enters the inguinal preperitoneal space, where takes the form of a dome and is fixed by four stitches
  Other Names: preperitoneal mesh

SUMMARY:
The investigators describe a new surgical technique for inguinal hernia open repair, which will be compared with the Lichtenstein technique. The investigators seek to find the difference between the two techniques in postoperative pain.

DETAILED DESCRIPTION:
The investigators randomly assigned 168 adult patients with uncomplicated primary inguinal hernia to two treatment groups:

Group A: 84 patients treated with the new technique Group B: 84 patients treated with the technique of Lichtenstein (gold standard) The investigators reviewed the patients operated on one week, one month, three months and six months after surgery. The investigators evaluated the presence of moderate to severe pain in each technique, as well as the intensity of pain, measured by visual analogue scale.

The investigators also determined the presence of inguinal dysesthesias in each technique, measured by dermatome mapping.

ELIGIBILITY:
Inclusion Criteria:

* adult patients diagnosed with uncomplicated primary inguinal hernia
* mentally healthy patients
* patients without preoperative groin pain
* patients eligible for outpatient surgery

Exclusion Criteria:

* patients with different surgical diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
pain one month after surgery | one month
  Pain will be measured by the Visual Analogue Scale, from zero to ten. Measurements will be made per month, three months and six months after surgery. With these data we will built two survival curves (one for each group)with the proportions of patients still have pain in every time frame. We will compare the two curves with logrank statistic test.
pain three months after surgery | three months
  Pain will be measured by the Visual Analogue Scale, from zero to ten. Measurements will be made per month, three months and six months after surgery. With these data we will built two survival curves (one for each group)with the proportions of patients still have pain in every time frame. We will compare the two curves with logrank statistic test.
pain six months after surgery | six months
  Pain will be measured by the Visual Analogue Scale, from zero to ten. Measurements will be made per month, three months and six months after surgery. With these data we will built two survival curves (one for each group)with the proportions of patients still have pain in every time frame. We will compare the two curves with logrank statistic test.

SECONDARY OUTCOMES:
dysesthesia one month after surgery | one month
  Inguinal dysesthesia will be measured by inguinal dermatome mapping, looking for anesthesia, hypoesthesia and hyperesthesia. Dysesthesias will be measured at one month, three months and six months. We dont know if there will be changes in dysesthesias over time but it is possible.
dysesthesia three months after surgery | three months
  Inguinal dysesthesia will be measured by inguinal dermatome mapping, looking for anesthesia, hypoesthesia and hyperesthesia. Dysesthesias will be measured at one month, three months and six months. We dont know if there will be changes in dysesthesias over time but it is possible.
dysesthesia six months after surgery | six months
  Inguinal dysesthesia will be measured by inguinal dermatome mapping, looking for anesthesia, hypoesthesia and hyperesthesia. Dysesthesias will be measured at one month, three months and six months. We dont know if there will be changes in dysesthesias over time but it is possible.

CONTACTS AND LOCATIONS:
Overall Officials: Rafal L Smolinski, surgeon, Principal Investigator — IMSS; Martha A Hernandez, researcher, Study Director — IMSS; Sergio E Solorio, researcher, Study Chair — IMSS
Locations (1):
- Ambulatory care medical unit number 55 (UMAA 55), León, Guanajuato, Mexico